CLINICAL TRIAL: NCT06330090
Title: Cognitive Dynamics in Early Childhood
Acronym: CODEC
Status: Recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL84688.091.23; 101040534 (Other Grant/Funding Number: European Research Council)
Record Dates: First submitted 2024-03-11; First posted 2024-03-26 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Change
Keywords: cognition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Design: Behavioural or behavioural with imaging

SUMMARY:
The goal of this accelerated longitudinal observational cohort study is to advance our understanding of cognitive variability in children aged 7 to 10 at first measurement. The CODEC study aims to integrate experience sampling methods, longitudinal designs, deep phenotyping cohorts, and state-of-the-art statistical methodologies to investigate three core questions:

1. How does cognitive variability differ between individuals?
2. What are the neural, psychological, and environmental mechanisms that underlie cognitive variability?
3. What are the long-term consequences and outcomes associated with differences in cognitive variability?

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in the behavioural arm of this study, a subject must meet all of the following criteria:

  * Between the ages of 7 and 10 years at the moment of the first assessment. In order to be eligible to participate in the imaging arm of this study, a subject must meet all of the following criteria:
  * Between the ages of 8 and 10 years at the moment of the first assessment.

Exclusion Criteria:

* A potential subject will be excluded from participation in the study if the participant indicates not understanding the instructions of the behavioural tasks due to a language barrier. In the imaging arm of the study, a potential subject who meets any of the following criteria will further be excluded from participation in the imaging arm of the study:

  * History of neurological or psychiatric illness.
  * History of using psychotropic medications.
  * Contraindications for MRI.
  * Metal parts that cannot be removed, are present in or on upper body, e.g. plates, screws, aneurysm clips, metal splinters, piercings or medical plasters. (exception: dental fillings, crowns, a metal wire behind the teeth, tattoos and contraceptive coils).
  * Body containing metal fragments, in particular in the eye, e.g., caused by injuries when working with metal.
  * History of brain surgery.
  * Active implant(s) (e.g. pacemaker, neurostimulator, insulin pump, ossicle prosthesis)
  * Using a medical plaster that cannot or may not be taken off (e.g. nicotine plaster)

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: 600 children will be recruited from schools and on individual bases to take part in the behavioural testing. A subgroup of 200 children will be further recruited to participate in the imaging part of the study at the Donders Institute.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Reaction times from the vocabulary cognitive task | Through study completion, an average of 3 years
  RT from accurate responses from the vocabulary task in the cognitive battery during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Reaction times from the exploration cognitive task | Through study completion, an average of 3 years
  RT from accurate responses from the exploration task in the cognitive battery during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Reaction times from the Working Memory cognitive task | Through study completion, an average of 3 years
  RT from accurate responses from the WM task in the cognitive battery during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Reaction times from the speed cognitive task | Through study completion, an average of 3 years
  RT from accurate responses from the speed raction time task in the cognitive battery during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Reaction times from the fluid reasoning cognitive task | Through study completion, an average of 3 years
  RT from accurate responses from the fluid reasoning task in the cognitive battery during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Mood score on smiley slider | Through study completion, an average of 3 years
  The current mood of the participant on a smiley slider from 0-100 during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
Sleep score on smiley slider | Through study completion, an average of 3 years
  The current level of tiredness of the participant on a smiley slider from 0-100 during burst assessment (3x a day, 5x a week) and up to 2 additional occasions per year.
MP-RAGE MRI sequence baseline | an average of 1 year
  Structural MP-RAGE MRI scan at baseline measurement
Functional MRI sequence of low time constraint reasoning task at baseline | an average of 1 year
  Functional MRI scan at baseline measurement when participants perform fluid reasoning task with low time contraint.
gaze direction during reasoning task at baseline | an average of 1 year
  gaze direction recording through eye-tracking at baseline measurement when participants perform fluid reasoning task.
pupil dilation during reasoning task at baseline | an average of 1 year
  pupil dilation recording through eye-tracking at baseline measurement when participants perform fluid reasoning task.
Naturalistic viewing fMRI at baseline | an average of 1 year
  Naturalistic viewing fMRI at baseline measurement.
Naturalistic viewing fMRI at follow-up | two years after baseline
  Naturalistic viewing fMRI at follow-up measurement.
Functional MRI sequence of high time constraint reasoning task at follow-up | two years after baseline
  Functional MRI scan at follow-up measurement when participants perform fluid reasoning task with high time contraint.
gaze direction during reasoning task at baseline at follow-up | two years after baseline
  gaze direction recording through eye-tracking at follow-up measurement when participants perform fluid reasoning task.
pupil dilation during reasoning task at baseline at follow-up | two years after baseline
  pupil dilation recording through eye-tracking at follow-up measurement when participants perform fluid reasoning task.
Functional MRI sequence of low time constraint reasoning task at follow-up | two years after baseline
  Functional MRI scan at follow-up measurement when participants perform fluid reasoning task with low time contraint.
Sparse MP2-Rage MRI sequence baseline | an average of 1 year
  Structural Sparse MP2-Rage MRI scan at baseline measurement
Diffusion weighted imaging MRI sequence baseline | an average of 1 year
  Diffusion weighted imaging MRI scan at baseline measurement
MP-RAGE MRI sequence follow up | two years after baseline
  Structural MP-RAGE MRI scan at follow up measurement
Sparse MP2-Rage MRI sequence follow up | two years after baseline
  Structural Sparse MP2-Rage MRI scan at follow up measurement
Diffusion weighted imaging MRI sequence follow up | two years after baseline
  Diffusion weighted imaging MRI scan at follow up measurement
Total score for Highly Sensitive Child scale at baseline | an average of 1 year
  Participant reported 12-item Dutch version of the HSC scale measured at baseline. Each item is scored on a scale from 1-strongly disagree to 7-strongly agree
Total score for Strengths and difficulties questionnaire at baseline | an average of 1 year
  Parent reported 25-item Dutch version of the SDQ measured at baseline. Each item is scored (0-not at all/only a little, 1-quite a lot, 2-a great deal)
Total score for BRIEF-2 questionnaire at baseline | an average of 1 year
  Parent reported Dutch version of the Behaviour Rating Inventory of Executive Function 2 measured at baseline.
Total score for BRIEF-2 questionnaire at follow-up | two years after baseline
  Parent reported Dutch version of the Behaviour Rating Inventory of Executive Function 2 measured at follow-up.
Total score for Strengths and difficulties questionnaire at follow-up | two years after baseline
  Parent reported 25-item Dutch version of the SDQ measured at follow-up. Each item is scored (0-not at all/only a little, 1-quite a lot, 2-a great deal)
Total score for Mind Excessively Wandering Scale scale at baseline | an average of 1 year
  Participant reported 12-item Dutch version of the MEWS scale measured at baseline. Each item is scored on a scale from 0 (not at all or rarely) to 3 (nearly all of the time or constantly)
Originality score for the Alternative Uses Tasks at baseline | an average of 1 year
  Originality score of responses on an alternative uses task at baseline.
Originality score for the Alternative Uses Tasks at follow-up | two years after baseline
  Originality score of responses on an alternative uses task at follow-up.
Total score for Parent-reported Mind Excessively Wandering Scale scale at baseline | an average of 1 year
  Parent reported 12-item Dutch version of the MEWS scale measured at baseline. Each item is scored on a scale from 0 (not at all or rarely) to 3 (nearly all of the time or constantly)
Total score for Parent-reported Socio-demographic questionnaire at baseline | an average of 1 year
  Parent reported socio-demograpic questionnaire at baseline. Total score on SES related questions (highest level of educationm professional situation) will be measured.
Total score for Parent-reported Socio-demographic questionnaire at follow-up | two years after baseline
  Parent reported socio-demograpic questionnaire at baseline. Total score on SES related questions (highest level of education, professional situation) will be measured.
Total score for Mind Excessively Wandering Scale scale at follow-up | two years after baseline
  Participant reported 12-item Dutch version of the MEWS scale measured at follow-up. Each item is scored on a scale from 0 (not at all or rarely) to 3 (nearly all of the time or constantly)
Total score for Parent-reported Mind Excessively Wandering Scale scale at follow-up | two years after baseline
  Parent reported 12-item Dutch version of the MEWS scale measured at follow-up. Each item is scored on a scale from 0 (not at all or rarely) to 3 (nearly all of the time or constantly)
Total score for Highly Sensitive Child scale at follow-up | two years after baseline
  Participant-reported 12-item Dutch version of the HSC scale measured at follow-up. Each item is scored on a scale from 1-strongly disagree to 7-strongly agree

SECONDARY OUTCOMES:
motivation rating for cognitive tasks | Through study completion, an average of 3 years
  Rating from least to most fun cognitive task once a year after completing the cognitie battery 10 times in the burst week
Decibel of background noise during cognitive testing | Through study completion, an average of 3 years
  DB recording of background noise when performing the cognitive tasks at the start of the testing
Academic school result baseline | an average of 1 year
  cito-scores, academic results on national test obtained through schools at baseline
Academic school result follow-up | two years after baseline
  cito-scores, academic results on national test obtained through schools at follow-up
Parent reaction times on cognitive battery at baseline | an average of 1 year
  Parents performed RT on accurate responses in measures on the complete cognitive battery (vocabulary, reasoning, exploration, working memory and speed) at baseline
Parent reaction times on cognitive battery at follow-up | two years after baseline
  Parents performed RT on accurate responses in measures on the complete cognitive battery (vocabulary, reasoning, exploration, working memory and speed) at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Radboudumc Department of Cognitive Neuroscience, Nijmegen, Netherlands

REFERENCES:
- [Derived] Coolen IEJI, van Langen J, Hofman S, van Aagten FE, Schaaf JV, Michel L, Aristodemou M, Judd N, van Hout ATB, Meeussen E, Kievit RA. Protocol and preregistration for the CODEC project: measuring, modelling and mechanistically understanding the nature of cognitive variability in early childhood. BMC Psychol. 2024 Jul 26;12(1):407. doi: 10.1186/s40359-024-01904-5. PMID 39060934